CLINICAL TRIAL: NCT02189733
Title: A Phase I, Single Center, Open-Label, Randomized, Single Dose Cross-Over Study in Healthy Male Subjects to Investigate the Bioequivalence and Tolerability of Liquid and Reconstituted Lyophilized Subcutaneous Formulations of Caplacizumab.
Brief Title: Bioequivalence of Liquid and Reconstituted Lyophilized Subcutaneous Formulations of Caplacizumab.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALX0681-C102; 2014-001294-13 (EudraCT Number)
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — caplacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caplacizumab - Treatment A (Experimental): Single s.c. dose of reconstituted lyophilized solution of caplacizumab followed by single s.c. dose of liquid formulation of caplacizumab
  Interventions: Biological: Caplacizumab
- Caplacizumab - Treatment B (Experimental): Single s.c. dose of liquid formulation of caplacizumab followed by single s.c. dose of reconstituted lyophilized solution of caplacizumab
  Interventions: Biological: Caplacizumab

INTERVENTIONS:
Biological: Caplacizumab — Comparison of reconstituted lyophilised formulation versus liquid formulation of caplacizumab

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetic characteristics and demonstrate bioequivalence of a reconstituted new lyophilized formulation of caplacizumab for subcutaneous (s.c.) injection as compared to an equal nominal s.c. dose of the reference liquid formulation of caplacizumab.

The secondary objective of the study is to compare the safety and tolerability, and the pharmacodynamic parameters of the new formulation with those of the reference formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasians aged 18 to 55 years, inclusive.
* Body weight 55 - 100 kg and body mass index (BMI) between 18.5 and 30.0, extremes included.
* Coagulation and bleeding diathesis variables (as defined in the protocol) within the normal range at screening and on Day -1.
* Others as defined in the protocol.

Exclusion Criteria:

* History or presence of diseases in the kidneys and/or heart, lungs, liver, skin, endocrine organs or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of and/or any sign or symptom indicating current abnormal hemostasis or blood dyscrasia.
* Others as defined in the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: concentration of caplacizumab in plasma | Day 1 (pre-dose) until Day 7

SECONDARY OUTCOMES:
Pharmacodynamics as measured by Ristocetin cofactor activity in plasma | During screening until day 29 +/-1
Safety and Tolerability: safety markers | From signing of informed consent form until day 43 +/- 2
  Adverse events, local tolerability, laboratory assessments, urinalysis, vital signs, 12-lead ECG, physical examinations
Pharmacodynamics as measured by von Willebrand factor antigen in plasma | During screening until Day 29 +/- 1
Pharmacodynamics as measured by Factor VIII clotting activity in plasma | During screening until day 29 +/- 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Paillarse, MD, Study Director — Ablynx, a Sanofi company
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom